CLINICAL TRIAL: NCT04324671
Title: a Study of the Pattern of Upper Airway Obstruction in Non-obese Patients With Snoring and Obstructive Sleep Apnea
Brief Title: Upper Airway Obstruction in Non-obese Patients With Snoring and Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Basma Khairy Mohamed, director, Assiut University
Other Study IDs: snoring in non-obese
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: nasofibroscopy — Flexible videorhinolaryngoscope, PAL 11101VP*, 4.2 mm diameter. Using a computerized system including:
  Light source: Explor ENT (HAL250). The software allowed audio, video recording and retrieval of recorded material.

SUMMARY:
This study aims at :-

1. detecting the prevelance of snoring and OSA in non-obese patients
2. identify their diagnostic profile in order to provide proper management

DETAILED DESCRIPTION:
Snoring is the vibration of respiratory structures and the resulting sound due to obstructed air movement during breathing while sleeping.

Snoring during sleep may be a sign, or first alarm, of obstructive sleep apnea (OSA).

Snoring can cause significant psychological and social problems to sufferers. Multiple studies reveal a positive correlation between loud snoring and risk of heart attack and stroke.

Obstructive sleep apnea (OSA) is the commonest type of sleep apnea and is characterized by inturpted snoring, repeated attacks of complete or partial pharyngeal closure during sleep despite the effort to breath resulting in nocturnal hypoxemia, frequent arousals during sleep, and excessive daytime sleepiness (EDS).

Obstructive Sleep Apnea is differentiated from Central Sleep Apnea (CSA) which is characterized by changes in the respiratory cycle during sleep but without the effort to breath during the apnea.

the episodes of decreased breathing are called "hypopnea " and it's definition requires a < 30% drop in flow for 10 seconds or longer associated with < 3% oxygen desaturation , the episodes of breathing cessations are called "apneas" and defined as a< 90% drop in flow for 10 seconds or longer and associated with < 3% oxygen desaturation or an arousal It is a serious and potentially life threatening disease that is far more common than generally expected. Several risk factors, including obesity, male sex, age, and heritable factors, as well as the supine decubitus position during sleep. have been associated with an increased prevalence of obstructive sleep apnea in the general population.

It has become a major health issue all over the world affecting quality of life with an increasing prevalence and associated with high comorbidities such as diabetes mellitus, hypertension, cardiovascular disease, dyslipidemia, malignancies, and overall mortality. Results of different studies indicate that approximately 60-70% of patients with OSA are obese.

Snoring and witnessed apnea are more frequent among men but insomnia for example is more frequent among women. The OSA frequency increase with age for the women. The mortality is higher for women The data regarding association of OSA among nonobese patients is rare and needs great effort as fewer studies have reported magnitude of association.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* patients complaining of snoring and obstructive sleep panea

Exclusion Criteria:

* chronic pulmonary disease ( COPD, Asthma ,IPF)
* Pregnancy
* sever cardiovascular disease ( unstable angina , sever arrhythmia , MI)
* chronic renal failure (CRF)
* neurological disorders

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients refaired to outpatient clinic of Phoniatric Unit, Assiut University Hospital in duration of 1 year with history of snoring and history suggestive of obstructive sleep apnea will be included in this study
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
compare snoring and obstructive sleep apnea between obese and non obese | baseline
  by analysing data of muller's manauver and sleep endoscopy between obese and nonobese

REFERENCES:
- [Background] Armstrong MW, Wallace CL, Marais J. The effect of surgery upon the quality of life in snoring patients and their partners: a between-subjects case-controlled trial. Clin Otolaryngol Allied Sci. 1999 Dec;24(6):510-22. doi: 10.1046/j.1365-2273.1999.00307.x. PMID 10606999
- [Background] Tung P, Levitzky YS, Wang R, Weng J, Quan SF, Gottlieb DJ, Rueschman M, Punjabi NM, Mehra R, Bertisch S, Benjamin EJ, Redline S. Obstructive and Central Sleep Apnea and the Risk of Incident Atrial Fibrillation in a Community Cohort of Men and Women. J Am Heart Assoc. 2017 Jul 1;6(7):e004500. doi: 10.1161/JAHA.116.004500. PMID 28668820
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376
- See also: Related Info — http://jtd.amegroups.com/article/view/17916/html